CLINICAL TRIAL: NCT05093010
Title: The Relationship Between Body Surface Gastric Mapping (BSGM) and Gastric Emptying Rate
Brief Title: The Relationship Between Body Surface Gastric Mapping and Gastric Emptying Rate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S65541
Record Dates: First submitted 2021-09-09; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Motility Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, a new generation of high-resolution electrogastrograms recording technology with 64-channel electrode array is being developed by Alimetry Limited. This BSGM provide a more complete understanding of the origin and propagation of human gastric slow-wave activity non-invasively, such as frequency, amplitude, velocity, and pattern, in high spatiotemporal detail. The system is also capable of providing a novel meal response metric, which might correlate with the gastric emptying time. The system includes an App for tracking patient-reported symptoms throughout the test.The aim of the present study is to assess and compare BSGM and breath-based gastric emptying parameters and to study the relation between BSGM and presence or severity of individual symptoms and clinical features.The investigators will perform a study in 100 subjects to record gastric bioelectrical activity by non-invasive multi-channel body-surface electrode arrays during gastric emptying breathing test.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old;
* Male or female patients;
* Patients planned GEBT;
* Negative PCR on nasopharyngeal swab 24 or 48 hours prior to the test;
* Signed informed consent.

Exclusion Criteria:

* Females who are pregnant or lactating.
* History of skin allergies or a history of extreme sensitivity to cosmetics or lotions
* Fragile skin vulnerable to skin tears.
* Damaged epigastric skin (open wounds, rash, inflammation)
* Patients unable to remain in a relaxed reclined position for the test duration

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who will receive gastric emptying breath test
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Validation of body surface gastric mapping for delayed gastric emptying | 30 minutes before the meal and 4 hours after having meal.
  The correlation of electrogastrography abnormality (in percentage) and delayed gastric emptying (t 1/2, minutes) will be determined employing a regression method.

SECONDARY OUTCOMES:
To assess correlation between electrogastrography abnormality and upper gastrointestinal symptoms. | 30 minutes before the meal and 4 hours after having meal.
  Visual analogue scale (VAS) score for gastrointestinal symptoms, including pain, nausea, vomiting, bloating and flatulence will be recoded during recording gastric electrophysiological activity. The correlation of electrogastrography abnormality (in percentage) and upper gastrointestinal symptoms severity will be determined employing a regression method.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carson DA, O'Grady G, Du P, Gharibans AA, Andrews CN. Body surface mapping of the stomach: New directions for clinically evaluating gastric electrical activity. Neurogastroenterol Motil. 2021 Mar;33(3):e14048. doi: 10.1111/nmo.14048. Epub 2020 Dec 4. PMID 33274564